CLINICAL TRIAL: NCT00942760
Title: DMS-0901: Multimodal Magnetic Resonance Protocol to Distinguish Tumor Recurrence From Treatment-Related Necrosis in Patients With High Grade Gliomas
Brief Title: Protocol to Distinguish Tumor Recurrence From Treatment-Related Necrosis in Patients With High Grade Gliomas
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: D0901; DMS-0901
Record Dates: First submitted 2009-07-20; First posted 2009-07-21 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2012-07

CONDITIONS: Recurrent High Grade Gliomas

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Research MRI: High Grade Glioma patients who show progression based on MRI
  Interventions: Device: 3T MRI

INTERVENTIONS:
Device: 3T MRI — The introduction of the 3T scanners provides a potential opportunity to improve the quality of imaging in neuro-oncology.

SUMMARY:
Brain imaging tests are routinely used to detect the presence of a brain tumor or to evaluate the response to treatment. Sometimes the images obtained are not specific and the only way to establish a diagnosis is by obtaining a tissue sample. The hypotheses of the study is to determine if multimodal MR technique will provide tissue signatures that differentiate between tumor progression and treatment related necrosis in high grade glioma patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven high grae glioma with central pathology review at DHMC
* Age 18 equal to or greater than 18 years
* Karnofsky performance greater or equal to 60%
* Patients must have received radiation therapy and chemotherapy but should not have received any anti-angiogenesis therapy.

Exclusion Criteria:

* Any patient who requires urgent surgical resection of MRI abnormality would not be eligible
* Pregnant women are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recurrent GBM patients
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2009-04; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To prospectively acquire multiparameter MR variables at 1.5T and 3T MRI from treated high grade glioma patients to assign tissue signatures for tumor recurrence and radiation necrosis as established by pathologic examination. | 24 months

SECONDARY OUTCOMES:
To compare the predictive values of the multiparameter MR tissue signatures acquired at 1.5T and 3T | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States